CLINICAL TRIAL: NCT02838719
Title: Effect of Perineural Versus Intravenous Dexamethasone On Analgesic Efficacy of Transverse Abdominis Plane Block With Levobupivacaine In Laparoscopic Gynaecological Procedures: A Randomized, Double-Blind Study
Brief Title: Analgesic Efficacy of Dexamethasone in Different Routes of Administration in Transverse Abdominis Plane Block
Acronym: AEDDATB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vetriselvan p, Junior Resident Anaesthesia, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PAIN86
Record Dates: First submitted 2016-05-26; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: INFERTILITY
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perineural group (Experimental): Group 1: perineural dexamethasone acetate added to bilateral transverse abdominis plane block with levobupivacaine
  Interventions: Drug: Perineural Dexamethasone acetate
- Intravenous group (Active Comparator): Group 2: Intravenous dexamethasone acetate added with bilateral transverse abdominal plane block with levobupivacaine
  Interventions: Drug: Intravenous dexamethasone acetate

INTERVENTIONS:
Drug: Perineural Dexamethasone acetate
  Other Names: Decoin
  Arms: Perineural group
Drug: Intravenous dexamethasone acetate
  Other Names: Decoin
  Arms: Intravenous group

SUMMARY:
Transverse abdominis plane (TAP) block is a regional anaesthesia technique that provides analgesia to the parietal peritoneum as well as skin and muscles of the anterior abdominal wall. In the past, a number of adjuvants have been added to the local anaesthetics in peripheral and neuraxial blocks resulting in an effective and long lasting analgesia.In recent times, dexamethasone has been increasingly used as an adjuvant to local anaesthetics in peripheral nerve blocks. Dexamethasone has a long and efficient glucocorticoid structure and also has anti-inflammatory property. It also blocks the C- fibers of pain pathway. When added to local anaesthetics as an adjuvant in peripheral nerve blocks, it has shown to prolong the analgesia time. A number of previous studies have also shown an opioid sparing effect of steroids, when used intravenously perioperatively. Though previous studies have shown that addition of dexamethasone to local anaesthetics in transverse abdominis plane block prolongs the duration of block, however it is not known whether this effect of dexamethasone is due to its peripheral action or because of its systemic absorption. Thus, in this study planned to compare the effectiveness of dexamethasone on quality and duration of analgesia when used as an adjuvant with local anaesthetics in transverse abdominis plane block versus when given systemically by intravenous route along with transverse abdominis plane block using local anaesthetics only, in patients undergoing gynaecological laparoscopic procedures under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 to 70 years undergoing gynaecological laparoscopic surgeries under general anaesthesia
2. ASA physical status1 or 2

Exclusion Criteria:

1. Local infection
2. Morbid obesity (body mass index >35kg/m2)
3. Allergy to local anaesthetics
4. Patient refusal
5. Severe respiratory or cardiac disorders
6. Pre-existing neurological deficits
7. Liver or renal insufficiency
8. Preexisting diabetics
9. Patient on steroid treatment for any reason.
10. Peri Operative use of steroids

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesic | first 24 hours
  Pain will be assessed by vas score, if vas score more than 3 rescue analgesia will be given. Duration between the end of anaesthesia to first analgesic requirement during first 24 hours of postoperative period.

SECONDARY OUTCOMES:
Total amount of rescue analgesic required in 1st 24 hours postoperatively | 0, 0.25, 0.50, 0.75, 1 , 2, 4, 6, 8,12, 24 hours
  Pain will be assessed by vas score, if vas score more than 3 rescue analgesia will be given.

IPD SHARING:
Plan to Share IPD: No